CLINICAL TRIAL: NCT02847741
Title: Predictive Nature of Total Cholesterol Threshold: Possible Link to Suicidal Behavior
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: UF 8921; 2011-A01657-34 (Other: Agence Nationale de Sécurité des Médicaments)
Record Dates: First submitted 2016-07-15; First posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Current Major Depressive Disorder
Keywords: Depression; Cholesterol; Suicidal behavior; Predictive factor
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Major depressive episode (Other): Depressive patients will be assessed by interview (psychiatrists), questionnaires and blood sampling, as the inpatients's routine care
  Interventions: Other: patient's routine care

INTERVENTIONS:
Other: patient's routine care — Interview by psychiatrists, questionnaires, blood analysis

SUMMARY:
Suicidal behavior (SB) is a public health problem. The clinical model currently admitted to the understanding of SB is a stress vulnerability model, but so far, all scientific works has no clinical application. The management of psychiatric patients, including depressed subjects, faces the inability to detect those with a high risk of SB. Many studies have shown a link between low cholesterol and SB. A study has recently proposed a total cholesterol threshold below which the risk of suicide could be increased. However, a prospective study is needed to assess the predictive nature of such an indicator.

DETAILED DESCRIPTION:
Investigators propose to assess, within a cohort of patients, the predictive value of a total cholesterol threshold in the occurrence of SB.

555 inpatients suffering from a current Major depressive disorder (MDD), hospitalized in the Department of Emergency Psychiatry and Post Acute Care will be recruited.

Each patient will attend a total of 5 visits during a follow-up period of 18 months (visits at 1, 3, 6, 12, and 18 months)

ELIGIBILITY:
Inclusion criteria:

* Major
* Meet the Diagnostic and Statistical Manual of Mental Disorders-IV (DSM) criteria for a major depressive episode
* Subject who signed the non-opposition form
* Able to understand the nature, purpose and methodology of the study
* Able to understand and perform the clinical and neuropsychological evaluations.

Exclusion criteria:

* Subject whose primary psychiatric diagnosis is not a major depressive episode according to DSM-IV criteria (the existence of psychiatric comorbidity is not a criterion for non-inclusion)
* Refusal of participation
* Subject Deprived of liberty (by judicial or administrative decision)
* Subject protected by law (guardianship)
* Subject exclusion period in relation to another protocol
* Subject for which the maximum annual amount of allowances of € 4,500 has been reached
* Subject not affiliated to a social security scheme or not being the beneficiary of such a scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2012-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
frequency of suicide attempts | at 18 month
  frequency of suicide attempts during the 18months follow-up, according to the total cholesterol threshold at baseline. The biological sampling is carried out after 12 hours of fasting.

SECONDARY OUTCOMES:
number of past SB | at 18 month
  Studying the relation between the number of past SB (assessed by the Columbia Suicide History Form) and the occurrence of new SB during the 18 months follow-up
moral pain | at 18 month
  Studying the relation between moral pain (assessed by Likert scale from 0 to 10) at baseline and the occurrence of new SB during the 18 months follow-up
physical pain | at 18 month
  Studying the relation between physical pain (assessed Likert scale from 0 to 10) at baseline and the occurrence of new SB during the 18 months follow-up
suicidal ideation | at 18 month
  Studying the relation between suicidal ideation (assessed by the Columbia Suicide Severity Rating Scale, the Scale of Suicidal Ideation) and the occurrence of new SB during the 18 months follow-up
depression (Quick Inventory of Depressive Symptomatology) | at 18 month
  Studying the relation between score to the Quick Inventory of Depressive Symptomatology and the occurrence of new SB during the 18 months follow-up
history of childhood abuse | at 18 month
  Studying the relation between an history of childhood abuse (assessed by the Childhood Trauma Questionnaire) and the occurrence of new SB during the 18 months follow-up
National Adult Reading Test score | at 18 month
  Studying the relation between NART score (assessment of intellectual level) and the occurrence of new SB during the 18 months follow-up
scores to California Verbal Learning Test | at 18 month
  Studying the relation between scores to California Verbal Learning Test (assessment of verbal memory) and the occurrence of SB during the 18 months follow-up
scores to Iowa Gambling Task Time frame: 18 months | at 18 month
  Studying the relation between scores to the Iowa Gambling Task (assessment of decision making) and the occurrence of new SB during the 18 months follow-up
score to the brixton test | at 18 month
  Studying the relation between score to the brixton test (assessment of mental flexibility) and the occurrence of SB during the 18 months follow-up
scores to verbal fluency | at 18 month
  Studying the relation between scores to verbal fluency and the occurrence of SB during the 18 months follow-up
scores to Reversal Learning Task | at 18 month
  Studying the relation between scores to Reversal learning task (assessment of decision making) and the occurrence of new SB during the 18 months follow-up
scores to the Attentional Stroop test | at 18 month
  Studying the relation between scores to Attentional Stroop test and the occurrence of new SB during the 18 months follow-up
relation between inflammatory markers and the occurrence of SB | at 18 month
  Studying the relation between inflammatory markers at baseline and the occurrence of new SB during the 18 months follow-
relation between thyroid function and the occurrence of SB | at 18 month
  Studying the relation between thyroid function at baseline and the occurrence of new SB during the 18 months follow-up
relation between lipid profile and the occurrence of SB | at 18 month
  Studying the relation between lipid profile at baseline and the occurrence of new SB during the 18 months follow-up
relation between pharmacological assays and the occurrence of SB | at 18 month
  Studying the relation between pharmacological assays at baseline and the occurrence of new SB during the 18 months follow-up
relation between the characteristic of the mood depressive disorder (unipolar or bipolar depression) and the predictive or vulnerability factors of SB | at 18 month
  Studying the potential specificity of predictive or vulnerability factors of SB depending on whether the diagnosis is unipolar or bipolar depression
the characteristic of past SB | at 18 month
  Studying the relation between the number and the lethality of past SB (assessed by the Columbia Suicide History Form, the Risk Rescue Rating Scale, the Suicidal Intent Scale ) and the response to antidepressant treatment during the 18 months follow-up
moral pain | at 18 month
  Studying the relation between moral pain (assessed by Likert scale from 0 to 10) at baseline and the response to antidepressant treatment during the 18 months follow-up
physical pain | at 18 month
  Studying the relation between physical pain (assessed by Likert scale from 0 to 10) at baseline and the response to antidepressant treatment during the 18 months follow-up
suicidal ideation | at 18 month
  Studying the relation between suicidal ideation (assessed by the Columbia Suicide Severity Rating Scale, the Scale of Suicidal Ideation) and the response to antidepressant treatment during the 18 months follow-up
depression level (Inventory of Depressive Symptomatology) | at 18 month
  Studying the relation between score to the Inventory Of Depressive Symptomatology and the response to antidepressant treatment during the 18 months follow-up
history of childhood abuse | at 18 month
  Studying the relation between an history of childhood abuse (assessed by the childhood trauma questionnaire) and the response to antidepressant treatment during the 18 months follow-up
National Adult Reading Test score ( NART) | at 18 month
  Studying the relation between NART score (assessment of intellectual level ) and the response to antidepressant treatment during the 18 months follow-up
scores to California Verbal Learning Test | at 18 month
  Studying the relation between scores to California Verbal Learning Test (assessment of verbal memory) and the response to antidepressant treatment during the 18 months follow-up
scores to Iowa Gambling Task | at 18 month
  Studying the relation between scores to Iowa Gambling Task (assessment of decision making) and the response to antidepressant treatment during the 18 months follow-up
score to the brixton test | at 18 month
  Studying the relation between score to the brixton test (assessment of mental flexibility) and the response to antidepressant treatment during the 18 months follow-up
verbal fluency | at 18 month
  Studying the relation between score to verbal fluency and the response to antidepressant treatment during the 18 months follow-up
scores to Reversal Learning Task | at 18 month
  Studying the relation between scores to Reversal learning task (assessment of decision making) and the response to antidepressant treatment during the 18 months follow-up
scores to the Attentional Stroop test | at 18 month
  Studying the relation between scores to Attentional Stroop test and the response to antidepressant treatment during the 18 months follow-up
relation between inflammatory markers and the response to antidepressant treatment | at 18 month
  Studying the relation between inflammatory markers at baseline and the response to antidepressant treatment during the 18 months follow-up
relation between thyroid function and the response to antidepressant treatment | at 18 month
  Studying the relation between thyroid function at baseline and the response to antidepressant treatment during the 18 months follow-up
relation between lipid profile and the response to antidepressant treatment | at 18 month
  Studying the relation between lipid profile at baseline and the response to antidepressant treatment during the 18 months follow-up
relation between pharmacological assays and the response to antidepressant treatment | at 18 month
  Studying the relation between pharmacological assays at baseline and t the response to antidepressant treatment during the 18 months follow-up
lethality of past SB | at 18 month
  Studying the relation between the lethality of past SB (assessed by the Columbia Suicide History Form) and the occurrence of new SB during the 18 months follow-up
Depression (Inventory of Depressive Symptomatology) | at 18 month
  Studying the relation between score to the Inventory Of Depressive Symptomatology and the occurrence of new SB during the 18 months follow-up
Depression (Beck Depression Inventory) | at 18 month
  Studying the relation between score to the Beck Depression Inventory and the occurrence of new SB during the 18 months follow-up
depression level (Beck depression Inventory) | at 18 month
  Studying the relation between score to the Beck depression Inventory and the response to antidepressant treatment during the 18 months follow-up
depression level (Quick Inventory of Depressive Symptomatology) | at 18 month
  Studying the relation between score to the Quick Inventory of Depressive Symptomatology and the response to antidepressant treatment during the 18 months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Montpelleir University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No